CLINICAL TRIAL: NCT05148325
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerance and Pharmacokinetics of BAT4706 Injection in Patients With Advanced Solid Tumors
Brief Title: Assessment of Safety ,Tolerance and Pharmacokinetics Clinical Efficacy With BAT4706 in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bio-Thera Solutions (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAT-4706-001-CR
Record Dates: First submitted 2021-11-03; First posted 2021-12-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumor; Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): First Phase: dose escalation study. It was divided into six dose groups: 0.1mg/kg, 0.3mg/kg, 0.5mg/kg ,1.0mg/kg, 3.0mg/kg and 10.0mg/kg. The safety, tolerability and pharmacokinetics of bat4706 injection were explored according to the 3 + 3 dose increasing mode. It is expected that 18-36 cases will be included in the group Second Phase: dose expansion study. After the completion of dose increment, 1-2 tolerated doses were selected for extended research on melanoma (20-40 cases), so as to provide recommended doses for subsequent clinical trials
  Interventions: Drug: BAT4706

INTERVENTIONS:
Drug: BAT4706 — The administration cycle was proposed to be 3 weeks (Q3W), i.e., 21 days in a cycle, and the first 4 cycles were administered on the first day of each cycle.

SUMMARY:
A Phase I Clinical Study to Evaluate the Safety, Tolerance and Pharmacokinetics of BAT4706 Injection in Patients With Advanced Solid Tumors.

DETAILED DESCRIPTION:
This study is a single center, open, dose increasing and dose expanding phase I clinical study. The dose increasing method of "3 + 3" is used to explore the safety, tolerance and PK characteristics of BAT4706 injection in patients with advanced solid tumors. After the completion of dose increment, 1-2 tolerated doses were selected for extended research on melanoma (20-40 cases), so as to provide recommended doses for subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years old (including boundary value), male or female;
* Voluntarily sign informed consent;
* Study population: advanced patients diagnosed by pathology and without effective standard treatment or standard treatment failure or standard treatment intolerance or refuse standard treatment.Patients with malignant solid tumors. (the extended study phase is mainly for patients with advanced melanoma);
* According to recist1.1 standard, there is at least one measurable tumor focus;
* ECOG score shall be 0 or 1;
* The investigator assessed the expected survival ≥ 12 weeks;
* Have sufficient organ and bone marrow functions as below:Blood routine (no blood transfusion, no hematopoietic stimulator, and no medication to correct blood count within 14 days prior to first dosing),Neutrophil absolute count (ANC) ≥1.5×109 /L, Platelet count ≥75×109/L, Hemoglobin ≥90g/L, Blood coagulation function Prothrombin time (PT) or International standardized ratio (INR) and activated partial thrombin time (APTT) ≤ 1.5×ULN, Liver function Total bilirubin (TBIL) ≤2×ULN ,Alanine aminotransferase (ALT), aspartate aminotransferase (AST) -- ≤3×ULN,Serum Creatinine ≤1.5×ULN ，renal function Serum creatinine clearance rate & GT; 60ml/min (Cockcroft-Gault formula, see appendix)
* Female patients with fertility must have negative serum pregnancy test during screening, and agree to take effective birth control / contraception to prevent pregnancy from the study period to 6 months after the last administration. Male patients must agree to take effective contraceptive methods from the study period to 6 months after the last administration.

Exclusion Criteria:

* Have received experimental drug treatment or participated in clinical research of medical devices within 4 weeks before the first administration of study drugs Research;
* Received chemotherapy, radiotherapy, Biological therapy, endocrine therapy, immunotherapy, and other anti-tumor treatments within 4 weeks before the first administration of the study drug, except: 1. Nitrosourea or mitomycin C within 6 weeks prior to the first use of the study drug. 2. Oral fluorouracil and small molecule targeted drugs within 2 weeks or 5 half lives,Whichever is longer, etc.). 3. Traditional Chinese medicine/traditional Chinese patent medicines with definite anti-tumor effect, and drugs with immunomodulatory effect (including but not limited to thymosin Interferons, interleukins, etc.) within 2 weeks prior to the first use of the study drug. 4. Palliative radiotherapy within 2 weeks prior to the first use of the study drug.
* Failure of CTLA-4 monoclonal antibody treatment in the past;
* Before the first administration of the study drug, the AE (ctcae5.0) caused by previous antitumor treatment was still > grade 1, hair loss and menstrual stimulation Except those with stable immune hypothyroidism controlled by hormone replacement therapy;
* Received interventional therapy and major surgery (such as craniotomy, thoracotomy or laparotomy) within 4 weeks before the first administration of the study drug;Surgery is defined here as grade 3 and 4 surgery;
* Have a history of organ transplantation;
* Central nervous system or meningeal metastasis;
* If other malignant tumors have been diagnosed in recent 5 years, or the previous malignant tumors have been cured for less than 5 years, the time of the first pathological diagnosis shall prevail Subject to. Except for radical skin basal cell carcinoma, cutaneous squamous cell carcinoma or in situ carcinoma, such as in situ breast cancer, Cervical carcinoma in situ);
* Patients with ocular melanoma;
* Patients with esophageal or gastric variceal bleeding in the past 6 months, or the investigator assessed the risk of bleeding;
* Serious cardiovascular disease occurred within 6 months before the first medication: the New York Heart Association rating (NYHA) is 2 Heart failure of grade and above, left ventricular ejection fraction (LVEF) < 50%, unstable arrhythmia or unstable heart Colic and uncontrollable hypertension (this protocol is defined as contraction after treatment despite optimal antihypertensive treatment Blood pressure > 150mmhg and / or diastolic blood pressure > 100mmhg, and the investigator's evaluation is of clinical significance);
* Patients with a history of autoimmune diseases; Had splenectomy or splenic irradiation;
* Drugs with immunomodulatory effect (e.g. thymosin, interferon, interleukin) were used within 2 weeks before the first administration of the study drug Hormone) or hormone (equivalent dose > prednisone 10mg / day);
* Untreated or under treatment tuberculosis patients, including but not limited to tuberculosis; Those who have received standardized anti-tuberculosis treatment and have been confirmed by researchers as cured can be included;
* Patients who have experienced severe infections within 4 weeks prior to the first medication use, including but not limited to infection complications requiring hospitalization, bacteremia, severe pneumonia, etc; Exclude patients with active infections before the first administration;
* Patients with a history of non infectious pneumonia requiring glucocorticoid treatment or current interstitial lung disease within one year before the first administration;
* Patients with uncontrolled or requiring drainage of pleural effusion, pericardial effusion, or abdominal effusion;
* Individuals with the following risks of thrombosis or bleeding:

  1. Have experienced myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack within 6 months before the first administration;
  2. A history of deep venous thrombosis, pulmonary embolism, or any other severe thromboembolism within 3 months prior to the first administration (implantable venous infusion port or catheter derived thrombosis, or superficial venous thrombosis is not considered "severe" thromboembolism);
  3. Any life-threatening bleeding event or grade 3 or 4 gastrointestinal/variceal bleeding event requiring blood transfusion, endoscopy, or surgical treatment within 3 months prior to the first administration;
  4. Investigator believe that other diseases with a higher risk of bleeding or thrombosis in the future
* Patients with active tuberculosis; Active infections requiring intravenous antibiotic treatment;
* People infected with the following diseases: human immunodeficiency virus (HIV) infection; Treponema pallidum antibody positive; hepatitis B virus Infected persons were positive for hepatitis B surface antigen (HBsAg) and hepatitis B virus deoxyribonucleic acid (HBV DNA) detection > 2000iu / ml (or 1 × 104 copies / ml); HCV infected persons [HCV antibody and disease];Viral RNA (HCV RNA) test results were positive];
* Inoculated within 4 weeks before the first medication, or planned to receive live / attenuated vaccine during the study period;
* Known hypersensitivity to any monoclonal antibody;
* Known history of psychotropic substance abuse or drug abuse;
* Pregnant or lactating women;
* Other patients considered by the investigator as unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Explore the maximum tolerated dose (MTD) | 21 days after first dosing
  To evaluate the safety and tolerance of BAT4706 injection in patients with advanced solid tumors, explore the maximum tolerated dose (MTD), and provide the recommended dose for subsequent clinical trials.

SECONDARY OUTCOMES:
Cmax | 126 days after first dosing
  Single dose PK characteristics
Tmax | 126 days after first dosing
  Single dose PK characteristics
T1/2 | 126 days after first dosing
  PK characteristics
CL | 126 days after first dosing
  Single dose PK characteristics
Vd | 126 days after first dosing
  Single dose PK characteristics
AUC(0-τ) | 126 days after first dosing
  Single dose PK characteristics
AUC(0-∞) | 126 days after first dosing
  Single dose PK characteristics
Cmax | 126 days after first dosing
  Multiple doses PK characteristics
Tmax | 126 days after first dosing
  Multiple doses PK characteristics
T1/2 | 126 days after first dosing
  Multiple doses PK characteristics
CL | 126 days after first dosing
  Multiple doses PK characteristics
MRT | 126 days after first dosing
  Multiple doses PK characteristics
DF | 126 days after first dosing
  Multiple doses PK characteristics
ADA antibody | 126 days after first dosing
  immunogenicity
Nab positive | 126 days after first dosing
  immunogenicity
ORR | 126 days after first dosing
  Tumor evaluation after administration will be performed at weeks 6, 12, and 18.
BORR | 126 days after first dosing
  Tumor evaluation after administration will be performed at weeks 6, 12, and 18.
DOR | 126 days after first dosing
  Tumor evaluation after administration will be performed at weeks 6, 12, and 18.
PFS | 126 days after first dosing
  Tumor evaluation after administration will be performed at weeks 6, 12, and 18.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, M.D, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing cancer hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No